CLINICAL TRIAL: NCT01395108
Title: Phase I Clinical Study on Oral Nemonoxacin Malate Capsules
Brief Title: Clinical Study on Oral Nemonoxacin Malate Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TaiGen Biotechnology Co., Ltd. (Industry)
Responsible Party: Yingyuan Zhang, Institute of Antibiotics, Huashan Hospital, Fundan University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG-873870-C-1
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — nemonoxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Nemonoxacin
- Nemonoxacin 125mg (Active Comparator): Nemonoxacin 125mg
  Interventions: Drug: Nemonoxacin
- Nemonoxacin 250mg (Active Comparator): Nemonoxacin 250mg
  Interventions: Drug: Nemonoxacin
- Nemonoxacin 500mg (Active Comparator): Nemonoxacin 500mg
  Interventions: Drug: Nemonoxacin
- Nemonoxacin 750mg (Active Comparator): Nemonoxacin 750mg
  Interventions: Drug: Nemonoxacin
- Nemonoxacin 1000mg (Active Comparator): Nemonoxacin 1000mg
  Interventions: Drug: Nemonoxacin

INTERVENTIONS:
Drug: Nemonoxacin — oral once daily
  Other Names: TG-873870

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of nemonoxacin in healthy Chinese volunteers.

DETAILED DESCRIPTION:
Single dose study: evaluate safety and tolerability of oral nemonoxacin 125 mg, 250mg, 500mg, 750mg, and 1000mg.

Multiple dose study: evaluate PK profile of oral doses of 500mg or 750mg nemo after consecutive 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, aged between 18 and 45 during screening
* Male volunteers who are capable of taking double-barrier contraception measures during the test (spermicide gel plus condom, for instance) until the end of the clinical study and do not cause their spouses to conceive within three months after the last administration of the medication; if the subjects are females, they shall not become pregnant during the test and within three months after the study
* No use of tobacco or nicotine product within 3 months prior to this study
* BMI 19-25
* Willing to abstain from coffee and any caffeine drink during the study
* Voluntarily sign the informed consent

Exclusion Criteria:

* History of diabetes, or cardiovascular, hepatic or renal disease
* Active digestive disease (e.g. diarrhea)
* Central nervous disease or psychiatric disorders
* Had surgery or trauma within 6 months prior to this study
* Alcohol or drug abuse
* HIV, HBV or HCV positive
* Used any prescribed drug (including traditional chinese medicine) within 14 days prior to the study
* Donated 400ml of blood or plasma within 3 months prior to this study
* Have an abnormal laboratory examination value that exceeds the normal range by 10%
* Drug allergies
* Have cardiac disorders or have a family history of cardiac disorders
* Have abnormal 12-lead ECG during screening
* Pregnant or lactating
* Participated in any study within 3 months prior to this study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated single oral dose of nemonoxacin in healthy Chinese volunteers | 7 days
Pharmacokinetic profile of single oral dose of nemonoxacin in healthy Chinese volunteers | 7 days
Pharmacokinetic profile of repeated oral doses of nemonoxacin in healthy Chinese volunteers | 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Yingyuan Zhang, PhD, Principal Investigator — Huashan Hospital, Fundan University
Locations (1):
- Institute of Antibiotics, Huashan Hospital, Fundan University, Shanghai, China

REFERENCES:
- [Derived] Guo B, Wu X, Zhang Y, Shi Y, Yu J, Cao G, Zhang J. Safety and clinical pharmacokinetics of nemonoxacin, a novel non-fluorinated quinolone, in healthy Chinese volunteers following single and multiple oral doses. Clin Drug Investig. 2012 Jul 1;32(7):475-86. doi: 10.2165/11632780-000000000-00000. PMID 22650326